CLINICAL TRIAL: NCT06902844
Title: A Study of Equecabtagene Autoleucel Injection (Eque-cel) in the Treatment of Relapsed/Refractory Systemic Lupus Erythematosus (SLE)
Brief Title: Equecabtagene Autoleucel Injection (Eque-cel) for Relapsed/Refractory Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lingli Dong, Principal Investigator, Director,Head of rheumatology department, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT103ACI002
Record Dates: First submitted 2025-03-05; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus (SLE); Lupus Nephritis (LN)
Keywords: CAR T; SLE; LN
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1.0 x 10^6 CAR+ T cells (Experimental): Experimental: Equecabtagene Autoleucel Injection （Eque-cel ） Drug:Equecabtagene Autoleucel Injection
  Interventions: Drug: Equecabtagene Autoleucel Injection

INTERVENTIONS:
Drug: Equecabtagene Autoleucel Injection — dosage form: injection, dosage: 1.0×10^6 CAR-T/kg, frequency: single dose.

SUMMARY:
This is a single-center, open-label, exploratory clinical study to evaluate the efficacy and safety of Equecabtagene Autoleucel Injection (Eque-cel) in patients with Relapsed /refractory systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
SLE is a chronic diffuse connective tissue disease with unexplained etiology that can involve multiple systems. SLE is considered as an incurable disease and traditional SLE treatment aims at long-term remission. Eque-cel is an autologous chimeric antigen receptor T-cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA), which expressed on both mature B lymphocytes and malignant plasma cells. BCMA CAR-T cells offer another potential therapeutic option to eliminate plasma cells in patients with SLE driven by abnormal antibody who still suffer recurrent attacks from conventional treatments. In this study subjects will receive a three-day consecutive lymphodepletion therapy, and 1.0×10^6 total CAR T cells/kg after enrollment. A follow-up phase will include assessments for safety, efficacy evaluation and pharmacokinetics monitoring. The duration of this trial is about 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old, male or female;
2. Subjects with relapsed/refractory SLE:

   1. Subjects must be diagnosed with SLE according to the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria, or the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria; the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥8, with a British Isles Lupus Assessment Group 2004 (BILAG-2004) activity score of A in ≥1 organ at screening, or a BILAG-2004 activity score of B in ≥2 organs.
   2. Subjects with lupus nephritis (LN) must be diagnosed with active, biopsy-confirmed lupus nephritis of type III, IV, or V, or type III/IV combined with type V according to the 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria; the SLEDAI-2000(SLEDAI-2K) score ≥8;
   3. Regular treatment with glucocorticoids and at least two immunosuppressants，immunomodulators, antimalarials, or biologics for at least 3 months, but withpoorly-controlled symptoms or intolerance to treatment.
3. Disease-related pathogenic antibody positive: anti-nuclear antibody (ANA) positive and/or anti-dsDNA positive and/or anti-Smith positive.
4. After signing the informed consent form, subjects and their partners must be willing to use effective and reliable method of contraception, devices or medicines, within one year post Eque-cel infusion (excluding contraception safety periods).
5. Subjects must provide written informed consent before the study begin.

Exclusion Criteria:

1. Disease involved the nervous system with a BILAG-2004 activity score of Class A.
2. History of solid organ transplantation.
3. History of autologous or allogeneic stem cell transplantation.
4. History of prior cell therapy or treatment of BCMA-targeted drug.
5. Known history of primary immunodeficiency (innate or acquired). 6）Concomitant other autoimmune diseases that may interfere with the study evaluation.

7) Subjects who have received the following drugs/non-drug treatment:

1. Subjects who have used therapeutic doses of corticosteroids (defined as >20 mg/day of prednisone or equivalent) within 1 week prior to enrollment. Corticosteroids must be tapered gradually according to clinical circumstances (e.g., duration and dose of treatment, severity of disease progression, and patient condition) before discontinuation，until reaching the allowable dose range specified in the protocol. Physiological replacement therapy, topical use, and inhaled corticosteroids are permitted.
2. Subjects who have used immunosuppressants other than corticosteroids within 1 week prior to enrollment.
3. Subjects who received biologic therapies or JAK/BTK/TYK inhibitors within 2 months prior to cell infusion, including but not limited to rituximab, belimumab, or baricitinib.
4. Subjects who underwent plasmapheresis or double filtration within 1 week prior to enrollment.
5. Subjects who received investigational drugs from another interventional clinical trial within 1 month before signing the informed consent form (ICF).
6. Subjects who received treatment of the study disease with any unlisted drugs within at least 5 half-lives prior to cell infusion.

   8)Major operation or surgical treatment caused by any reason that occurred or was planned within 4 weeks before enrollment or within 12 weeks after cell infusion.

   9)History of psychoactive drug abuse and failed to withdraw, or have a history of psychiatric disorders.

   10)Subjects have uncontrolled active fungal, viral, bacterial, or other infections (with persistent infection-related signs/symptoms that have not improvedafter appropriate anti-infective therapy) or infections requiring intravenous anti-infective therapy.

   11)Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with abnormal peripheral blood hepatitis B virus (HBV) DNA (defined as HBV DNA ≥100 IU/mL or ≥1000 copies/mL or above the normal reference range of the testing center, or positive qualitative HBV DNA); positive for hepatitis C virus (HCV) antibody with detectable peripheral blood HCV RNA (defined as ≥1000 IU/mL); positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA (defined as ≥1000 IU/mL); or positive for Treponema pallidum-specific antibody with positive rapid plasma reagin (RPR) test.

   12)Blood tests: Absolute neutrophil count < 1×10^9 /L, or Absolute lymphocyte count < 0.3×10 ^ 9 /L, or hemoglobin <60 g/L。 13)Subjects with serious cardiac disease: including but not limited to unstable angina and/or myocardial infarction within 12 months before screening, any congestive heart failure (New York Heart Association[NYHA] classification ≥Grade III), and a history of severe arrhythmias; or left ventricular ejection fraction (LVEF) <45%.

   14)Subjects with severe asthma or chronic obstructive pulmonary disease (COPD). Mild or moderate asthma or COPD under stable treatment may be considered with approval from the investigator and sponsor; orarterial oxygen saturation <91% at rest.

   15）Subjects have a significant risk of severe bleeding assessed by investigator.

   16) Subjects have a severe hepatic insufficiency assessed by investigator. 17) History of severe renal disease; or an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m² calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

   18) History of acute cerebrovascular events, including transient ischemic attack or stroke, within 6 months prior to enrollment.

   19) Any severe and/or uncontrolled comorbid conditions that, in the investigator's opinion, may interfere with the study evaluation.

   20) Diagnosis of malignancy within 5 years prior to screening, except for cured cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, ductal carcinoma in situ of the breast after radical surgery, or papillary thyroid carcinoma.

   21) Known history of severe allergy to any component of the eque-cel injection. 22）Pregnant or lactating women. 23) Subjects with other conditions adjudicated by the investigator as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Response rate of SRI-4 at 6 months after Eque-cel infusion | 6 months post Eque-cel infusion.
  SLE Responder Index (SRI)-4 is defined as follows with all criteria compared to Baseline:
  * ≥ 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score.
  * No worsening of the overall condition (< 0.3 point increase in Physician's Global Assessment [PhGA]) .
  * No new British Isles Lupus Assessment Group (BILAG) A or more than 1 new BILAG B disease activity scores.

SECONDARY OUTCOMES:
lupus low disease activity state (LLDAS) rate through 2 years after Eque-cel infusion | up to 2 years from Eque-cel infusion
  Proportions of subjects achieving LLDAS by timepoint;
Definitions of Remission in SLE (DORIS) rate through 2 years after Eque-cel infusion | up to 2 years from Eque-cel infusion
  Proportions of subjects achieving remission according to the DORIS as assessed by SLEDAI-2K Scale，PhGA Scale and concomitant medication usage.
Complete and Partial Renal Response（Lupus Nephritis Patients）through 2 years after Eque-cel infusion | up to 2 years from Eque-cel infusion
  Proportion of Participants Who Achieve Overall Complete and Partial Renal Response (CRR+PRR).
Safety Endpoint -Adverse Events（AEs） | up to 2 years from Eque-cel infusion
  Type and incidence of AEs as Assessed by CTCAE 5.0 (except CRS and ICANS assessed according to the criteria of NCI-CTCAE v5.0).
Pharmacokinetic Endpoint-Cmax | up to 2 years from Eque-cel infusion
  The maximum concentration (Cmax) of CAR VCN in peripheral blood after CAR-T infusion.
Pharmacokinetic Endpoint-Tmax | up to 2 years from Eque-cel infusion
  the time for CAR VCN to reach the maximum concentration (Tmax) after CAR-T infusion.
Pharmacokinetic Endpoint-AUC | up to 2 years from Eque-cel infusion
  Area under the curve of 28, 90 days and the last time point of PK detection (AUC0-28d, AUC0-90d, AUC0-last) for CAR VCN.
Pharmacokinetic Endpoint-Cmax | up to 90 days from Eque-cel infusion
  The maximum concentration (Cmax) of BCMA CAR-T in peripheral blood after CAR-T infusion.
Pharmacokinetic Endpoint-Tmax | up to 90 days from Eque-cel infusion
  the time for BCMA CAR-T to reach the maximum concentration (Tmax) after CAR-T infusion.
Pharmacokinetic Endpoint-AUC | up to 90 days from Eque-cel infusion
  Area under the curve of 28 days, 90 days (AUC0-28d, AUC0-90) for BCMA CAR-T.
Pharmacodynamic Endpoint- pathogenic antibodies | up to 2 years from Eque-cel infusion
  Changes in serum levels of pathogenic antibodies such as ANA, anti-dsDNA, and anti-Smith.
Pharmacodynamic Endpoint- Complement levels | up to 2 years from Eque-cel infusion
  Changes in measures of C3, C4.
Pharmacodynamic Endpoint-sBCMA | up to 2 years from Eque-cel infusion
  The concentration of soluble BCMA in peripheral blood of experimental group at each time point.

OTHER OUTCOMES:
Immunogenicity | up to 2 years from Eque-cel infusion
  Presence of human anti-CAR antibodies, and titer of confirmed positive antibody in peripheral blood.
C-reactive protein (CRP) | up to 2 years from Eque-cel infusion
  Changes in the levels of CRP.
Ferritin | up to 2 years from Eque-cel infusion
  Changes in the levels of Ferritin.
Interleukin-6 (IL-6) | up to 2 years from Eque-cel infusion
  Changes in the levels of IL-6.
replication competent lentivirus (RCL) | up to 2 years from Eque-cel infusion
  The incidence of replication competent lentivirus.
Immune cell subsets | up to 2 years from Eque-cel infusion
  Changes in the levels of Immune cell subsets.
Exploratory Endpoint：TCR repertoire and Gene Expression Profile | up to 2 years from Eque-cel infusion
  Changes in clonal expansion and diversity of TCR repertoire assessed by single cell sequencing.
Exploratory Endpoint： BCR repertoire and Gene Expression Profile | up to 2 years from Eque-cel infusion
  Changes in clonal expansion and diversity of BCR repertoire assessed by single cell sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol
Access Criteria: upon reasonable request